CLINICAL TRIAL: NCT02818621
Title: Does Administration of Dexmedetomidine Guided by Entropy/SPI Reduce the Requirement of Propofol and Remifentanil as Well as Increase the Quality of Recovery Profile?
Brief Title: Administration of Dexmedetomidine Guided by Entropy/SPI Reduce
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jiwon An, Associate Porfessor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3-2014-0218
Record Dates: First submitted 2016-06-23; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Dex (Active Comparator): The Dex group received 1mcg/kg loading dose followed by 0.5mcg/kg/hr infusion of dexmedetomidine which was administered at induction of anesthesia through skin closure.
  Interventions:
  ◦Drug: Dexmedetomidine
  Interventions: Drug: Group Dex (dexmedetomidine)
- Group Placebo (Placebo Comparator): The Placebo group received equal amount of normal saline.
  Interventions:
  ◦Drug: Normal saline
  Interventions: Drug: Group Dex (dexmedetomidine)

INTERVENTIONS:
Drug: Group Dex (dexmedetomidine) — 1mcg/kg loading dose followed by 0.5mcg/kg/hr infusion of dexmedetomidine which was administered at induction of anesthesia through skin closure
  Other Names: Precedex

SUMMARY:
Dexmedetomidine, a selective alpha2-adrenergic agonist is known to reduce propofol and opioid requirements due to its sedative and analgesic properties. However, until now, there has been studies based on indirect measures such as hemodynamics. Entropy shows to quantify the level of consciousness by EEG and Surgical pleth index(SPI) allows to predict the effect of pain stimuli and analgesic therapy by the index of the nociception-anti-nociception balance. The investigators analyzed quantitatively the requirements of propofol and remifentanil under continuous infusion of dexmedetomidine when using entropy and SPI.

DETAILED DESCRIPTION:
Dexmedetomidine, a selective alpha2-adrenergic agonist is known to reduce propofol and opioid requirements due to its sedative and analgesic properties. However, until now, there has been studies based on indirect measures such as hemodynamics. Entropy shows to quantify the level of consciousness by EEG and Surgical pleth index(SPI) allows to predict the effect of pain stimuli and analgesic therapy by the index of the nociception-anti-nociception balance. The investigators analyzed quantitatively the requirements of propofol and remifentanil under continuous infusion of dexmedetomidine when using entropy and SPI.

Patients (20~65 years old, ASA class 1 or 2) scheduled lumbar discectomy under general anesthesia were recruited. The patients were randomly allocated to two groups. Both groups received Target controlled infusion(TCI) of propofol and remifentanil and the dexmedetomidine was added to the Dex group and normal saline was added to the Placebo group. The Dex group received 1mcg/kg loading dose followed by 0.5mcg/kg/hr infusion of dexmedetomidine which was administered at induction of anesthesia through skin closure. The placebo group received equal amount of normal saline. During maintenance of anesthesia the effect site concentration of propofol and remifentanil was titrated to maintain Entropy(SE) 40~60 and SPI under 50. Blood pressure and heart rate also was measured. The total amount of propofol and remifentanil administered, time between eye opening and extubation was recorded. The quality of recovery was evaluated by QoR-40 survey after 24 hours postop.

ELIGIBILITY:
Inclusion Criteria:

1.The patients (20~65 years old, ASA class 1 or 2) scheduled lumbar discectomy under general anesthesia

Exclusion Criteria:

1. ASA class (American Society of Anesthesiologist physical status classification) 3 or higher
2. Patients with history of allergy or side effects on propofol, remifentanil, dexmedetomidine
3. BMI (body mass index) higher than 35
4. Patients taking monoamine oxidase inhibitor or adrenergic blocking agent
5. Pregnancy, Emergency operation
6. Patients with liver disease, cognitive dysfunction or drug abuse history

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The difference of the requirements of propofol and remifentanil between each groups | the day of surgery
  We analyzed quantitatively the requirements of propofol and remifentanil under continuous infusion of dexmedetomidine or placebo(normal saline) when using entropy and SPI.

SECONDARY OUTCOMES:
The difference of quality of recovery between each groups | 24 hours after surgery
  The quality of recovery was evaluated by QoR-40 survey after 24 hours postop.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, PhD, Study Chair — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No